CLINICAL TRIAL: NCT04101344
Title: Effect of Dietary Supplementation With Fiber Blends on the Gut Microbiota and Host Metabolome and Proteome
Brief Title: Fiber Blends and Gut Microbiota (FB)
Acronym: FB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201907041
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Gut Microbiome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fiber-blend (Experimental): All participants will receive a two fiber-blend snack and then a four fiber-blend snack. Stool, blood, and urine will be monitored for changes throughout the study.
  Interventions: Other: Two fiber-blend snack and four fiber-blend snack

INTERVENTIONS:
Other: Two fiber-blend snack and four fiber-blend snack — All subjects will complete a 47-day, multi-phase feeding study to evaluate the effect of two snack prototypes containing two different fiber blends on gut community structure and features of host biological state (plasma proteome/ metabolome).

SUMMARY:
The purpose of this research study is to determine whether consuming snacks containing different blends of dietary fibers alters the type and number of bacteria found in your gut and improves markers of overall health.

DETAILED DESCRIPTION:
All subjects will complete a 47-day, multi-phase feeding study to evaluate the effect of two snack prototypes containing two different fiber blends on gut community structure and features of host biological state (plasma proteome/ metabolome). The information gained from this work will increase our understanding of the importance of specific dietary fibers in manipulating the composition of the gut microbiota in ways that may improve our metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥25.0 and ≤35.0 kg/m2
* ≥18 and ≤60 years

Exclusion Criteria:

* previous bariatric surgery
* significant organ system dysfunction (e.g., diabetes, severe pulmonary, kidney, liver or cardiovascular disease)
* cancer or cancer that has been in remission for <5 years
* major psychiatric illness
* inflammatory gastrointestinal disease
* pregnant or lactating women
* use of medications that are known to affect the study outcome measures and that cannot be temporarily discontinued for this study
* use of medications known to affect the composition of the gut microbiota within the last 30 days (most notably antibiotics)
* bowel movements <3 times per week
* vegans, vegetarians, those with lactose intolerance and/or severe allergies/aversions/sensitivities to foods and ingredients included in the prescribed meal plan
* persons who are not able to grant voluntary informed consent
* persons who are unable or unwilling to follow the study protocol or who, for any reason, the research team considers not an appropriate candidate for this study, including non-compliance with screening appointments or study visits.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Effect of fiber blend snacks on gut microbiota | 1 year
  Stool samples will be analyzed to determine changes in type and number of gut microbiota.

SECONDARY OUTCOMES:
Effect of fiber blend snacks in blood and urine | 1 year
  Blood and urine samples will be analyzed to assess how many proteins and metabolites are present in these samples before and after fiber snack supplementation.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided